CLINICAL TRIAL: NCT06433609
Title: A Phase II Study of Antibody-Drug Conjugates (ADCs) Combined With Adebrelimab in HER2-negative Advanced Breast Cancer
Brief Title: Study of ADCs Combined With Adebrelimab in HER2-negative Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Yang Ke, Associate chief physician, Beijing GoBroad Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-008; BC-MUL-IIT-ADC-SHR1316 (Other: Jiangsu Hengrui Pharmaceuticals Co., Ltd.)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811+adebrelimab (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Adebrelimab
- SHR-A1921+adebrelimab (Experimental)
  Interventions: Drug: SHR-A1921; Drug: Adebrelimab

INTERVENTIONS:
Drug: SHR-A1811 — Via intravenous infusion
  Arms: SHR-A1811+adebrelimab
Drug: SHR-A1921 — Via intravenous infusion
  Arms: SHR-A1921+adebrelimab
Drug: Adebrelimab — Via intravenous infusion

SUMMARY:
Our study is aimed to evaluate the efficacy and safety of novel ADCs named SHR-A1811 and SHR-A1921 combined with adebrelimab in HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 75 years old (including boundary values), female patients with breast cancer;
2. ECOG PS Score: 0~1;
3. Histologically or cytologically confirmed HER2-negative advanced breast cancer;
4. Disease progression after prior 1-2 lines of systemic therapy; if HR-positive, prior CDK4/6 inhibitor is necessary;
5. Based on RECIST v1.1, at least one measurable lesion;
6. Brain metastasis with no clinical symptoms, or treated, stable brain metastases are eligible;
7. No prior PD-(L)1 inhibitor;
8. Patients must have a life expectancy ≥ 6 months;
9. Adequate organ function and marrow function (no corrective treatment within 14 days before first dose);
10. Patients of childbearing potential should have a negative urine or serum pregnancy, and must promise to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy or be celibate;
11. Available blood samples for ctDNA detection in the exploratory study;
12. Willing and able to provide written informed consent and comply with the requirements and restrictions in the protocol.

Exclusion Criteria:

1. Has known active brain metastasis which needs local therapy immediately;
2. Prior anti-HER2 or anti-TROP-2 treatment;
3. Has received or been receiving PD-(L)1 inhibitors and/or ADC containing a topoisomerase inhibitor-like payload;
4. Existence of third space fluid that is not well controlled by effective methods, e.g. drainage;
5. Has received antitumor surgery, radiotherapy, chemotherapy, targeted therapy or immunological therapy within 4 weeks before first dose of study therapy; has received antitumor endocrine therapy within one week before first dose of study therapy;
6. Use of other antitumor systemic treatment during the study;
7. Has active autoimmune disease or a history of autoimmune disease;
8. Known history of immunodeficiency, including HIV-positive, other acquired or innate immunodeficient disease, or known history of organ transplantation;
9. Has active hepatitis B (HBsAg-positive and HBV DNA≥500 IU/mL), hepatitis C (positive for HCV antibody and HCV RNA above ULN) and hepatic cirrhosis;
10. Has an active infection requiring antibiotics, antiviral or antifungal treatment, or pyrexia >38.5℃ of unknown origin during the screening period before first dose of study therapy (patients with pyrexia due to cancer could be enrolled determined by investigator);
11. Receiving immunosuppressive medication, or systemic corticosteroid therapy for the purpose of immunosuppression (prednisone at >10mg/d or equivalent dose of other corticosteroids), and continuous use within 2 weeks before the first dose of study therapy;
12. Other malignancy within prior 5 years unless curatively treated with no evidence of disease for at least recent 3 years, except: curatively treated in situ cancer of the cervix, skin basal cell carcinoma or skin squamous cell carcinoma;
13. Hypersensitivity to study therapy or any of its excipients;
14. Has known clinically significant lung disease, including but not limited to: interstitial lung disease, pneumonitis, pulmonary fibrosis;
15. Known history of uncontrolled cardiovascular clinical symptom or disease that is not well controlled;
16. Has received a live vaccine within 4 weeks before first dose of study therapy, or potential to receive a live vaccine during the trial treatment;
17. Patients with a positive serum or urine pregnancy test or who are breastfeeding; patients of childbearing potential who are unwilling or not available to use an effective method of contraception;
18. Other conditions that might influence the study and analysis of results in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
ORR (objective response rate) by investigator | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3.5 years
  ORR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1.

SECONDARY OUTCOMES:
DCR (disease control rate) by investigator | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3.5 years
  DCR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1.
CBR (clinical benefit rate) by investigator | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3.5 years
  CBR is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD lasting≥24 weeks (stable disease) per RECIST v1.1.
DoR (duration of response) | up to 3.5 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS (progression-free survival) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3.5 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS (overall survival) | up to 3.5 years
  OS is the time from the date of first dose until the date of death by any cause.
Safety as assessed by percentage of patients with any Adverse Event (AE) | up to 3.5 years
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Ke, Principal Investigator — Beijing GoBroad Hospital
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No